CLINICAL TRIAL: NCT00499980
Title: A Prospective Pilot Clinical Trial Evaluating the Utility of a Dynamic Near Infrared Imaging Device for Characterizing Suspicious Breast Lesions
Brief Title: Near Infrared/ Ultrasound Dual Modal Imaging for Breast Cancer Diagnosis
Acronym: NIR
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: ViOptix Canada (Industry)
Other Study IDs: OSU-04117
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2007-07-12 (Estimated); Status verified 2007-07

CONDITIONS: Breast Neoplasms
Keywords: Breast cancer; Spectroscopy, Near-Infrared; Oximetry
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate a dynamic near infrared imaging device for characterizing suspicious breast lesions

DETAILED DESCRIPTION:
Breast cancer is the leading cause of cancer among women in the United States. It has always been the hope that devising methods of earlier detection would lead to improvement of long-term survival. Therefore, the development of novel, more selective, and noninvasive diagnostic techniques is a priority. Mammography is currently the most commonly used breast imaging modality for both screening and diagnostic purposes. Additionally, breast ultrasound imaging and breast magnetic resonance imaging (MRI) are generally used to supplement or help confirm any indeterminate or suspicious finding prior to consideration of a breast biopsy. However, these conventional imaging methods lack information about tissue function and have lower diagnostic accuracy.

Most recently, near infrared (NIR, of wavelength 700-900 nm) optical diffuse spectroscopic imaging has been investigated as a novel diagnostic tool for breast cancer. In the near-infrared (NIR) light spectrum, oxygenated hemoglobin and deoxygenated hemoglobin are the major chromospheres in tissue, and the absorption spectrums of the two hemoglobin states differ across these wavelengths. Thus, there have been many contemporary attempts to use the intra-tissue absorption and scattering of NIR light to quantify functional tissue parameters such as hemoglobin concentration (HbT) and oxygen saturation (StO2), including tumor differentiation within the human breast. To a very good approximation, NIR photons diffuse through relatively thick tissues, such as several centimeters of a human breast. Functional imaging with NIR light offers several novel tissue parameters that differentiate tumors from normal breast tissue. For example, hemoglobin de-saturation in tumors may be increased due to the high oxygen demand of cancers and blood volume may be increased over that of normal background tissue due to the greater vascularization and metabolic needs of cancers.

While NIR imaging provides additional physiological parameters that potentially help to improve the specificity of breast cancer diagnosis, its relatively low spatial resolution makes it unsuitable for morphological analysis. The resolution of a NIR system is intrinsically limited by the diffusive nature of the near infrared light in tissue. Currently, typical instruments can distinguish simple structures of approximately 1 cm in size; sharp edges are typically blurred by a few millimeters. It was proposed that the imaging technique combining near infrared and ultrasound modalities has the potential to fully utilize their complementary features and overcome their deficiencies. This protocol defines the clinical study to prove the concept of the near infrared/ ultrasound dual modal imaging and to evaluate its sensitivity and specificity for breast cancer diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Non-pregnant (as defined by previous tubal ligation, no menses for last 12 consecutive months, or a negative quantitative serum pregnancy test on the day of the procedure.)
* Age: 18 years or older
* Suspicious lesion (BIRAD 4 or 5) identified by mammography and/or by ultrasound.
* A breast biopsy has been scheduled
* The suspicious lesion size is between 0.5 cm and 2 cm.
* The suspicious lesion depth is less than 3 cm from skin surface.
* The suspicious lesion should be clearly evident by ultrasound imaging

Exclusion Criteria:

* Patient with the biopsy performed to the suspicious lesion in the past 2 months on the same breast will be excluded from the study
* Patient with tattoos overlying the area of the suspicious lesion will be excluded from the study
* Patients with prior breast radiation therapy will be excluded from the study
* Patients with prior breast reduction surgery or breast augmentation surgery to the same breast will be excluded from the study
* Patients with previous surgical biopsy at or near the site of the suspicious lesion will be excluded from the study
* Patients with prior history of breast cancer in the same breast will be excluded from the study
* Patient who does not sign the consent form will be excluded from the study
* Patients that have not completed all studies of mammography and/or clinical ultrasound, P-Scan, Terason ultrasound and biopsy will be excluded from this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-03; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald X Xu, PhD, Principal Investigator — Department of Biomedical Engineering, OSU
Locations (1):
- JamesCare Breast Health Center, Dublin, Ohio, United States